CLINICAL TRIAL: NCT01036594
Title: An Endocrinologically and Pharmacologically Directed Trial of Ketoconazole and Corticosteroids in Castration Resistant Prostate Cancer
Brief Title: Ketoconazole and Dexamethasone in Prostate Cancer
Acronym: Keto/Dex
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 09553; NCI-2011-01263 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2009-12-17; First posted 2009-12-21 (Estimated); Results first posted 2020-06-29 (Actual); Last update posted 2020-06-29 (Actual); Status verified 2020-06

CONDITIONS: Prostate Cancer
Keywords: Ketoconazole; Dexamethasone
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Ketoconazole; Hydrocortisone; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ketoconazole + Hydrocortisone (Experimental): po = oral tid = 3 times per day qam = every morning qom = every evening bid = twice daily
  1 cycle = 28 days
  * Ketoconazole: 200mg during first week of study (run-in phase), then 400mg po tid
  * Hydrocortisone 20mg po qam and 10mg po qpm: If participant has ≥ 30% Prostate-specific antigen (PSA) decline at 12 week evaluation, treatment continues until progressive disease (by RECIST criteria OR by Prostate Specific Antigen Working Group (PSAWG) criteria) is documented. After that, drug will be discontinued. If participant has < 30% PSA decline at 12 week evaluation, participant goes off study.
  Interventions: Drug: Ketoconazole; Drug: Hydrocortisone
- Ketoconazole + Dexamethasone (Experimental): * Ketoconazole: 400mg po tid
  * Dexamethasone 0.5mg po bid: If ≥ 30% PSA decline (Prostate-specific antigen) at 12 week evaluation, administration starts when disease progression (by RECIST criteria OR by PSAWG criteria) is documented.
  Interventions: Drug: Ketoconazole; Drug: Dexamethasone

INTERVENTIONS:
Drug: Ketoconazole — 200mg during first week of study (run-in phase), then 400mg po tid
  Other Names: Ketoconazole Oral
Drug: Hydrocortisone — Hydrocortisone 20mg po qam and 10mg po qpm
  If participant has ≥30% PSA decline at 12 week evaluation, treatment continues until progressive disease (by RECIST criteria OR by PSAWG criteria) is documented. After that, drug will be discontinued. If participant has <30% PSA decline, patient goes off study.
  Arms: Ketoconazole + Hydrocortisone
Drug: Dexamethasone — Dexamethasone 0.5mg po bid
  If ≥ 30% PSA decline (Prostate-specific antigen) at 12 week evaluation, administration starts when disease progression (by RECIST criteria OR by PSAWG criteria) is documented.
  Other Names: Dexamethasone Oral
  Arms: Ketoconazole + Dexamethasone

SUMMARY:
This is an open label, phase II, single center trial of ketoconazole/dexamethasone to determine if the administration of ketoconazole/dexamethasone, after disease progression with ketoconazole/hydrocortisone slows or reverses disease progression in men with progressive prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate.
* Testosterone < 50 ng/dL. Participants must continue primary androgen deprivation with an luteinizing hormone-releasing hormone (LHRH) analogue if they have not undergone orchiectomy.
* Progressive non-metastatic or metastatic disease after androgen deprivation. Participants must have EITHER:

  1. Progression as defined by RECIST criteria. OR
  2. Progressive PSA documented within 4 weeks of enrollment. PSA evidence for progressive prostate cancer consists of a PSA level of at least 5 ng/ml which has risen on at least 2 successive occasions, at least 2 weeks apart. If the confirmatory PSA value is less than the first documented rising PSA value, then an additional test for rising PSA will be required to document progression.
* Participants who are receiving an antiandrogen as part of primary androgen ablation must demonstrate disease progression following discontinuation of antiandrogen.

  1. Disease progression after antiandrogen withdrawal is defined as 2 consecutive rising PSA values, obtained at least 2 weeks apart, or documented osseous or soft tissue progression.
  2. For participants receiving flutamide, at least one of the PSA values must be obtained 4 weeks or more after flutamide discontinuation.
  3. For participants receiving bicalutamide (Casodex) or nilutamide, at least one of the PSA values must be obtained 6 weeks or more after antiandrogen discontinuation.
* Karnofsky Performance Status ≥ 60%.
* Participants receiving any other hormonal therapy, including any dose of megestrol acetate (Megace), Proscar (finasteride), any herbal product known to decrease PSA levels (e.g., Saw Palmetto and PC-SPES), or any systemic corticosteroid must discontinue the agent for at least 4 weeks prior to enrollment.
* Participants on stable doses of bisphosphonates may continue on this medication; further, patients may initiate bisphosphonate therapy at the time of ketoconazole initiation.
* Prior radiation therapy completed ≥ 4 weeks prior to enrollment.
* Liver function tests (alanine aminotransferase (ALT), aspartate aminotransferase (AST), and Bilirubin) must be within normal limits.
* Absolute Neutrophil Count (ANC) >1500/µl, Platelet count > 100,00/µl, Creatinine <1.5 x upper limit of normal (ULN), Hemoglobin > 8 mg/dl.

Exclusion Criteria:

* Prior chemotherapy for prostate cancer is not allowed with the exception of cases in which chemotherapy has been administered in a neoadjuvant or adjuvant fashion AND >1 year has elapsed since the administration of this therapy.
* No prior ketoconazole, abiraterone, aminoglutethimide or corticosteroids for treatment of progressive prostate cancer.
* No supplements or complementary medicines/botanicals are permitted while on protocol therapy, except for any combination of the following: (conventional multivitamin supplements, selenium, lycopene, soy supplements) No prior radiopharmaceuticals (strontium, samarium) within 8 weeks prior to enrollment.
* No "currently active" second malignancy, other than non-melanoma skin cancer.
* No serious intercurrent infections or nonmalignant medical illnesses that are uncontrolled.
* No psychiatric illnesses/social situations that would limit compliance
* No active or uncontrolled autoimmune disease.
* No adrenal insufficiency as demonstrated by a baseline adrenocorticotropic hormone (ACTH) stimulation test demonstrating a peak cortisol >18 µg/dL.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-12-11 (Actual); Primary Completion 2012-12-11 (Actual); Study Completion 2014-10-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terence Friedlander, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through the Urologic Oncology Program at University of California, San Francisco
Pre-assignment Details: All participants were prescribed ketoconazole for a 7 day run-in phase, then hydrocortisone + ketoconazole treatment. Participants not achieving >=30% PSA decline at 12 weeks were taken off study. Participants continued treatment until progression at which time, hydrocortisone was discontinued and ketoconazole + dexamethasone treatment began.
Groups:
- Ketoconazole + Hydrocortisone: po = oral, tid = 3 times per day, qam = every morning, qom = every evening, bid = twice daily, 1 cycle = 28 days
  * Ketoconazole: 200mg during run-in phase, then 400mg po tid
  * Hydrocortisone 20mg po qam and 10mg po qpm: If participant has ≥ 30% PSA decline at 12 week evaluation, treatment continues until progressive disease (by RECIST criteria OR by Prostate Specific Antigen Working Group (PSAWG) criteria) is documented. After that, drug will be discontinued. If participant has < 30% PSA decline at 12 week evaluation, participant goes off study.
- Ketoconazole + Dexamethasone: Ketoconazole: 400mg po tid Dexamethasone 0.5mg po bid: If ≥ 30% PSA decline (Prostate-specific antigen) at 12 week evaluation, administration starts when disease progression on Ketoconazole + Hydrocortisone (by RECIST criteria OR by PSAWG criteria) is documented.
Period: Run-In: Ketoconazole Only (200 mg)
Arm/Group | Ketoconazole + Hydrocortisone | Ketoconazole + Dexamethasone
Started | 32 | 0 (Dexamethasone not introduced as treatment option until after Week 12 evaluation)
Completed | 31 | 0
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: First Treatment Regimen
Arm/Group | Ketoconazole + Hydrocortisone | Ketoconazole + Dexamethasone
Started | 31 | 0 (Dexamethasone not introduced as treatment option until after Week 12 evaluation)
Completed | 30 | 0
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Week 12 Evaluation
Arm/Group | Ketoconazole + Hydrocortisone | Ketoconazole + Dexamethasone
Started | 30 | 0 (Dexamethasone not introduced as treatment option until after Week 12 evaluation)
Completed | 24 | 0
Not Completed | 6 | 0
Not completed — Adverse Event | 5 | 0
Not completed — Physician Decision | 1 | 0
Period: Treatment Regiments Post Week 12
Arm/Group | Ketoconazole + Hydrocortisone | Ketoconazole + Dexamethasone
Started | 15 | 9
Completed | 13 | 5
Not Completed | 2 | 4
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Non-Cancer Disease Complications | 0 | 1
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Population: This is a sequential treatment design. Participants enrolled in first treatment regimen (Ketoconazole + Hydrocortisone) continued on 1st regimen based on disease status at week 12 evaluation and progression status. At progression, a second treatment option was assigned based on response to 1st regimen. 9 of the 32 total were assigned to 2nd regimen
Groups:
- All Patients Who Received Treatment: po = oral, tid = 3 times per day, qam = every morning, qom = every evening, bid = twice daily, 1 cycle = 28 days
  * Ketoconazole: 200mg during first week of study (run-in phase), then 400mg po tid
  * Hydrocortisone 20mg po qam and 10mg po qpm: If patient has ≥ 30% PSA decline at 12 week evaluation, treatment continues until progressive disease (by RECIST criteria OR by PSAWG criteria) is documented. After that, drug will be discontinued. If participant has < 30% PSA decline at 12 week evaluation, participant goes off study.
  Based on the results of evaluation at 12 weeks , participants were offered to either stay on this regimen or receive
  -Ketoconazole: 400mg po tid Dexamethasone 0.5mg po bid: If ≥ 30% PSA decline (Prostate-specific antigen) at 12 week evaluation, administration starts when disease progression on Ketoconazole + Hydrocortisone (by RECIST criteria OR by PSAWG criteria) is documented.
Arm/Group | All Patients Who Received Treatment
Number analyzed (Participants) | 32
Age, Customized [Count of Participants; unit: Participants]
  50-59 years old | 7
  60-69 years old | 11
  70-79 years old | 10
  80-89 years old | 4
Age, Customized [Count of Participants; unit: Participants] — Population: This measure presents data for the 9 participants that were subsequently randomized to the second treatment arm
  Participants
    50-59 years: number analyzed (Participants) | 9
    50-59 years | 1
    60-69 years: number analyzed (Participants) | 9
    60-69 years | 6
    70-79 years: number analyzed (Participants) | 9
    70-79 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: This measure presents data for the participants that were subsequently randomized to the second treatment arm
  Participants
    number analyzed (Participants) | 9
    Hispanic or Latino | 2
    Not Hispanic or Latino | 6
    Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 26
  More than one race | 0
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: This measure presents data for the participants that were subsequently randomized to the second treatment arm
  Participants
    number analyzed (Participants) | 9
    American Indian or Alaska Native | 0
    Asian | 3
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 1
    White | 5
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Achieved a Second Decline in Prostate Specific Antigen (PSA) Following Progression on First Regimen
Description: The number of participants who experience a ≥30% decline in PSA between the time of first progression on ketoconazole and hydrocortisone and eight weeks after dexamethasone therapy was initiated.
Time Frame: Up to 5 years
Population: Progression data for patients not enrolled to Dexamethasone arm are not used in this analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Ketoconazole + Hydrocortisone: po = oral, tid = 3 times per day, qam = every morning, qom = every evening, bid = twice daily, 1 cycle = 28 days
  * Ketoconazole: 200mg during first week of study (run-in phase), then 400mg po tid
  * Hydrocortisone 20mg po qam and 10mg po qpm: If patient has ≥ 30% PSA decline at 12 week evaluation, treatment continues until progressive disease (by RECIST criteria OR by PSAWG criteria) is documented. After that, drug will be discontinued. If patient has < 30% PSA decline at 12 week evaluation, patient goes off study.
Arm/Group | Ketoconazole + Hydrocortisone | Ketoconazole + Dexamethasone
Number analyzed (Participants) | 0 | 8
Participants |  | 0

2. Secondary Outcome: Median Change Over Time in Adrenocorticotrophic Hormone (ACTH) Levels for Participants Taking Ketoconazole/Hydrocortisone
Description: Nonparametric Wilcoxon test for matched pairs will be used to test the difference in ACTH levels from baseline until the time of disease progression for participants taking ketoconazole/hydrocortisone for participants with evaluable laboratory values.
Time Frame: Up to 5 years
Population: ACTH data not collected for this endpoint. Planned statistical analysis could not be performed.
Arm/Group | Ketoconazole + Hydrocortisone | Ketoconazole + Dexamethasone
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Relationship of ACTH to the Duration of Castration Prior to Treatment With Ketoconazole/Hydrocortisone and With Response
Description: The Spearman rank correlation will be calculated to explore the relationship between the baseline ACTH level and the duration of castration prior to the start of any ketoconazole therapy
Time Frame: Up to 2 years
Population: Data on duration of castration prior to treatment data not collected. Planned analysis could not be performed.
Arm/Group | Ketoconazole + Hydrocortisone | Ketoconazole + Dexamethasone
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Testosterone Levels Over Time for Participants on Dexamethasone
Description: For PSA responders to ketoconazole/ hydrocortisone continuing with dexamethasone treatment after initial disease progression, the overall pattern of testosterone levels will be investigated with nonparametric methods for statistical analyses. This will include Friedman's analysis of variance method using ranks for repeated measures. A key comparison using the Wilcoxon test for matched pairs will investigate the change in testosterone from progression #1 to progression #2.
Time Frame: Up to 5 years
Population: Testosterone data for this endpoint not collected. Planned statistical analysis could not be performed.
Arm/Group | Ketoconazole + Hydrocortisone | Ketoconazole + Dexamethasone
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Estrodiol Levels Over Time for Participants on Dexamethasone
Description: For PSA responders to ketoconazole/ hydrocortisone continuing with dexamethasone treatment after initial disease progression, the overall pattern of estrodiol levels will be investigated with nonparametric methods for statistical analyses. This will include Friedman's analysis of variance method using ranks for repeated measures. A key comparison using the Wilcoxon test for matched pairs will investigate the change in estrodiol from progression #1 to progression #2.
Time Frame: Up to 5 years
Population: Estrodiol data for this endpoint not collected. Planned statistical analysis could not be performed.
Arm/Group | Ketoconazole + Hydrocortisone | Ketoconazole + Dexamethasone
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Serum Adrenal Androgen (AA) Levels Over Time for Participants on Dexamethasone Over Time
Description: For PSA responders to ketoconazole/ hydrocortisone continuing with dexamethasone treatment after initial disease progression, the overall pattern of AA levels will be investigated with nonparametric methods for statistical analyses. This will include Friedman's analysis of variance method using ranks for repeated measures. A key comparison using the Wilcoxon test for matched pairs will investigate the change in AA levels from progression #1 to progression #2.
Time Frame: Up to 5 years
Population: AA data not collected for this endpoint. Planned statistical analyses could not be performed.
Arm/Group | Ketoconazole + Hydrocortisone | Ketoconazole + Dexamethasone
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Cortisol Levels Over Time for Participants on Dexamethasone Over Time
Description: For PSA responders to ketoconazole/ hydrocortisone continuing with dexamethasone treatment after initial disease progression, the overall pattern of cortisol levels will be investigated with nonparametric methods for statistical analyses. This will include Friedman's analysis of variance method using ranks for repeated measures. A key comparison using the Wilcoxon test for matched pairs will investigate the change in cortisol levels from progression #1 to progression #2.
Time Frame: Up to 5 years
Population: Cortisol data not collected for this endpoint. Planned statistical analysis could not be performed
Arm/Group | Ketoconazole + Hydrocortisone | Ketoconazole + Dexamethasone
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in Dehydroepiandrosterone (DHEA) Levels Over Time for Participants on Dexamethasone Over Time
Description: For PSA responders to ketoconazole/ hydrocortisone continuing with dexamethasone treatment after initial disease progression, the overall pattern of DHEA levels will be investigated with nonparametric methods for statistical analyses. This will include Friedman's analysis of variance method using ranks for repeated measures. A key comparison using the Wilcoxon test for matched pairs will investigate the change in DHEA levels from progression #1 to progression #2.
Time Frame: Up to 5 years
Population: DHEA data was not collected for this endpoint. Planned statistical analysis could not be performed.
Arm/Group | Ketoconazole + Hydrocortisone | Ketoconazole + Dexamethasone
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change in Dehydroepiandrosterone Sulfate (DHEA-S) Levels Over Time for Participants on Dexamethasone Over Time
Description: For PSA responders to ketoconazole/ hydrocortisone continuing with dexamethasone treatment after initial disease progression, the overall pattern of DHEA-S levels will be investigated with nonparametric methods for statistical analyses. This will include Friedman's analysis of variance method using ranks for repeated measures. A key comparison using the Wilcoxon test for matched pairs will investigate the change in DHEA-S levels from progression #1 to progression #2.
Time Frame: Up to 5 years
Population: DHEA-S data was not collected for this endpoint. Planned statistical analysis could not be performed.
Arm/Group | Ketoconazole + Hydrocortisone | Ketoconazole + Dexamethasone
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | Ketoconazole + Hydrocortisone | Ketoconazole + Dexamethasone
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/9
Serious Adverse Events (participants affected / at risk) | 4/32 | 0/9
Other Adverse Events (participants affected / at risk) | 25/32 | 5/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketoconazole + Hydrocortisone (N=32) | Ketoconazole + Dexamethasone (N=9)
Dehydration (Gastrointestinal disorders) | 1 (1) | 0 (0)
Peripheral arterial ischemia (Vascular disorders) | 1 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (2) | 0 (0)
Obstruction, GU - Ureter (Renal and urinary disorders) | 1 (1) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Infection with unknown ANC - Bladder (urinary) (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils - Upper airway NOS (Infections and infestations) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils - Bladder (urinary) (Infections and infestations) | 1 (1) | 0 (0)
Infection - Other (Infections and infestations) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ketoconazole + Hydrocortisone (N=32) | Ketoconazole + Dexamethasone (N=9)
Dermatology - Other (Skin and subcutaneous tissue disorders) | 8 (17) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (13) | 0 (0)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Rash: dermatitis associated with radiation - Radiation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (9) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1)
Anorexia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 3 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 12 (23) | 2 (2)
Insomnia (General disorders) | 2 (3) | 1 (1)
Weight gain (General disorders) | 1 (1) | 1 (2)
Weight loss (General disorders) | 1 (1) | 1 (2)
Edema: limb (General disorders) | 7 (14) | 2 (2)
ALT, SGPT (serum glutamic pyruvic transaminase) increased (Investigations) | 5 (15) | 1 (1)
AST, SGOT(serum glutamic oxaloacetic transaminase) increased (Investigations) | 6 (9) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Creatinine increased (Investigations) | 2 (3) | 0 (0)
Abdomen Pain, NOS (Gastrointestinal disorders) | 4 (8) | 0 (0)
Pain - Back (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Pain - Joint (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2)
Pain - Other (General disorders) | 3 (3) | 0 (0)
Pain - Chest/thorax NOS (General disorders) | 2 (3) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4 (8) | 0 (0)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Urinary frequency/urgency (Renal and urinary disorders) | 5 (6) | 0 (0)
Renal/Genitourinary (Renal and urinary disorders) | 2 (3) | 1 (1)
Perforation, GU - Kidney (Renal and urinary disorders) | 0 (0) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Skin (cellulitis) (Infections and infestations) | 1 (1) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung (pneumonia) (Infections and infestations) | 0 (0) | 1 (1)
Infection with unknown ANC - Joint (Infections and infestations) | 0 (0) | 1 (1)
Mood alteration - Depression (Psychiatric disorders) | 2 (2) | 2 (2)
Cognitive disturbance (Nervous system disorders) | 2 (2) | 0 (0)
Syncope (fainting) (Nervous system disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 5 (11) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2)
Joint-effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cardiac Arrhythmia - Other (Cardiac disorders) | 2 (3) | 0 (0)
Supraventricular and nodal arrhythmia - Sinus bradycardia (Cardiac disorders) | 2 (3) | 0 (0)
Cushingoid appearance (e.g., moon face, buffalo hump, centripetal obesity, cutaneous striae) (Endocrine disorders) | 2 (2) | 2 (2)
Peripheral arterial ischemia (Vascular disorders) | 2 (2) | 0 (0)
Thrombotic thrombocytopenic purpura [TTP] or hemolytic uremic syndrome [HUS] (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hepatobiliary/Pancreas - Other (Hepatobiliary disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Sample size and data collection for evaluable endpoints insufficient to complete planned analyses

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes